CLINICAL TRIAL: NCT02389413
Title: A Phase 2A Multicentre, Randomised, Double Blind, Placebo-Controlled, Parallel-Group Safety and Tolerability Study of PQ912 in Subjects With Early Alzheimer's Disease
Brief Title: Safety and Tolerability of PQ912 in Subjects With Early Alzheimer's Disease
Acronym: SAPHIR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vivoryon Therapeutics N.V. (Industry)
Collaborators: Julius Clinical (Industry); Amsterdam UMC, location VUmc (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PBD01071; 2014-001967-11 (EudraCT Number)
Record Dates: First submitted 2015-03-05; First posted 2015-03-17 (Estimated); Last update posted 2017-06-01 (Actual); Status verified 2017-01

CONDITIONS: Alzheimer's Disease
Keywords: PQ912; Glutaminy Cyclase (QC); QC - Inhibitor
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PQ912 oral (Experimental): PQ912 will be administered orally twice daily for 12 weeks.
  Interventions: Drug: PQ912 oral
- Placebo (Placebo Comparator): Placebo will be administered orally twice daily for 12 weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: PQ912 oral
  Arms: PQ912 oral
Other: Placebo
  Arms: Placebo

SUMMARY:
The aim of this study is to evaluate the safety, tolerability and preliminary efficacy of PQ912 in subjects with Mild Cognitive Impairment (MCI) due to Alzheimers Disease (AD) or mild dementia due to AD.

ELIGIBILITY:
Major Inclusion Criteria:

* Signed and dated written informed consent
* Male or surgically sterile or postmenopausal female aged ≥ 50 to ≤ 89 years. Male subjects with childbearing potential partners are willing to and should use condoms during treatment and until 28 days of the last dose of study medication.
* Diagnosis of MCI due to AD or mild dementia due to AD with amnestic presentation, according to AA-NIA (Alzheimer's Association (AA) and the National Institute on (Aging NIA) criteria [Albert et al 2011; McKhann et al 2011]
* Mini-Mental State Examination (MMSE) score of 21 to 30 inclusive at screening
* A positive AD signature showing one of the following (either a, b, c, OR d):

  1. Screening CSF sample with an A-beta 42 concentration of less than 638 ng/L AND total tau >375 ng/L, as assessed by central laboratory.
  2. Screening CSF sample with an A-beta 42 concentration of less than 638 ng/L AND p-tau > 52 ng/L, as assessed by central laboratory.
  3. Tau/A-beta ratio > 0.52, as assessed by central laboratory.
  4. A positive amyloid PET if available prior to screening.
* Treatment naïve, this means not having received any prior established specific treatment for MCI due to AD or mild dementia due to AD including no (prior) use of an acetylcholinesterase inhibitor or memantine. A maximum of two months of prior cumulative treatment with an acetylcholinesterase inhibitor or memantine is allowed if the acetylcholinesterase inhibitor or memantine was discontinued due to intolerance, and if this was done at least two months prior to baseline. Use of Souvenaid will be allowed if Souvenaid was discontinued at least twomonths prior to baseline, or if the subject is on stable dose for at least six months prior to baseline and is willing to continue during the study on the same dose and frequency.
* Outpatient with study partner capable of accompanying the subject on all clinic visits. In accordance to Swedish regulations availability of study partner is not applicable for Sweden.

Major Exclusion Criteria:

* Significant neurologic disease, other than AD, that may affect cognition.
* Atypical clinical presentations of MCI due to AD or mild dementia due to AD, such as the visual variant of AD (including posterior cortical atrophy) or the language variant (including logopenic aphasia).
* Concomitant disorders:

  * Severe hepatic (Child-Pugh C) and/or kidney failure (creatinine clearance (estimated Glomerular Filtration Rate - eGFR) ≤ 30 ml/min/1.73m2) and/or serum creatinine above 1.5 fold of Upper Limit Normal (ULN) and/or Alanine-Amino Transferase (AST) or Asparagine-Amino Transferase (ALT) above 3 fold ULN at baseline.
  * History of or screening visit brain MRI scan indicative of any other significant abnormality.
  * Current presence of a clinically important major psychiatric disorder (e.g. major depressive disorder) as defined by DSM-5 criteria, or symptom(s) (e.g. hallucinations) that could affect the subject's ability to complete the study.
  * . Current clinically important systemic illness that is likely to result in clinically relevant deterioration of the subject's condition or might affect the subject's safety during the study.
  * Other clinically important diseases or conditions or abnormalities of vital signs, physical examination, neurologic examination, laboratory results, or electrocardiogram (ECG) examination (e.g. atrial fibrillation) that could compromise the study or the safety of the subject.
  * Clinically important infection within 30 days prior to screening e.g. chronic persistent or acute infection, such as bronchitis or urinary tract infection.
  * Any known hypersensitivity to any of the excipients contained in the test article formulation.
  * Severe hepatic failure (Child-Pugh C) OR kidney failure (creatinine clearance (eGFR) ≤ 30 ml/min/1.73m2) OR serum creatinine above 1.5 fold of ULN OR AST or ALT above 3 fold of ULN at screening.´
* Concomitant Medication/Therapies:

The following therapies are not permitted for the given intervals prior to baseline and until End-of-treatment (EOT):

* Use of experimental medications for AD or any other investigational medications or devices for treatment of indications other than AD within 60 days prior to baseline.
* Treatment with Souvenaid, except if the use of Souvenaid was discontinued at least two months prior to baseline, or if the subject is on stable dose for at least six months prior to baseline and is willing to continue the use of Souvenaid during the study on the same dose and frequency.
* Concomitant treatment with St. John's Wort (a wash out phase of at least two weeks prior to baseline is required).
* Any concomitant treatment which impairs cognitive function and cannot be washed out at least four weeks prior to baseline.

Ages: 50 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2015-03; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Frequency of adverse events and serious adverse events (the study is a Phase II safety trial) | 12 weeks

SECONDARY OUTCOMES:
Exploratory clinical measures (measured by a questionnaire) | 12 weeks
  Mini-Mental State Examination (MMSE) Letter Fluency Test (LFT) Category Fluency Test (CFT) Geriatric Depression Scale (GDS) Cogstate Neuropsychological Test Battery
Change from baseline of a panel of concept and AD-related biomarkers in Cerebrospinal fluid (CSF) (measured by Analysis of several biochemical assays) | 12 weeks
  QC activity, total-tau, phospho-tau, Abeta pattern, pro-inflammatory panel
Change from baseline in brain functional connectivity (measured by Magnetic Resonance Imaging (MRI) analysis) | 12 weeks
Change from baseline in functional connectivity and network Analysis in electroencephalography (EEG) | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Frank Weber, Dr., Study Director — Vivoryon Therapeutics N.V.; Philip Scheltens, Prof. Dr., Study Chair — VUmc Alzheimer Centre (p: +31 20 4440816)
Locations (23):
- Ziekenhuis Netwerk Antwerpen / Geheugenkliniek, Hoboken, Belgium
- Finland (3):
  - Kliininen tutkimuskeskus, Kuopio
  - Oulu University Hospital, Oulu
  - CRST Oy, Turku
- France (4):
  - CHU Bordeaux Pellegrin (CMRR), Bordeaux
  - CHU François Mitterand (Centre Mémoire Ressources Recherche (CMRR)), Dijon
  - CHRU de Lille / Hôpital Roger Salengro, Lille
  - Hôpital La Grave / Centre de Recherche Clinique, Toulouse
- Germany (9):
  - Charité - Universitätsmedizin Berlin, Berlin
  - Universitätsmedizin Göttingen / Klinik für Psychiatrie und Psychotherapie, Göttingen
  - Universitätsklinikum Halle (Saale) Klinik und Poliklinik für Psychiatrie, Psychotherapie und Psychosomatik, Halle
  - Arzneimittelforschung Leipzig GmbH, Leipzig
  - Universitätsklinikum Magdeburg / Institut für Kognitive Neurologie und Demenzforschung, Magdeburg
  - Klinikum rechts der Isar der TU München / Klinik für Psychiatrie und Psychotherapie, München
  - Universitätsklinikum Münster / Klinik für Allgemeine Neurologie, Münster
  - Universitätsmedizin Rostock / Zentrum für Nervenheilkunde/ Klinik für Psychosomatik und Psychotherapeutische Medizin, Rostock
  - Neurologische Universitätsklinik Ulm, Ulm
- Alzheimer Research Center, Amsterdam, Netherlands
- Spain (4):
  - Hospital de la Santa Creu i Sant Pau, Neurology Department, Memory Unit, Barcelona
  - Fundació ACE. Institut Català de Neurociències Aplicades, Barcelona
  - Complexo Hospitalario Universitario de Santiago (CHUS), Santiago de Compostela
  - Hospital Universitario Virgen Macarena, Seville
- Verksamheten för neuropsykiatri Sahlgrenska universitetssjukhuset, Mölndal, Sweden

REFERENCES:
- [Derived] Scheltens P, Hallikainen M, Grimmer T, Duning T, Gouw AA, Teunissen CE, Wink AM, Maruff P, Harrison J, van Baal CM, Bruins S, Lues I, Prins ND. Safety, tolerability and efficacy of the glutaminyl cyclase inhibitor PQ912 in Alzheimer's disease: results of a randomized, double-blind, placebo-controlled phase 2a study. Alzheimers Res Ther. 2018 Oct 12;10(1):107. doi: 10.1186/s13195-018-0431-6. PMID 30309389